CLINICAL TRIAL: NCT06734039
Title: Impact of Anatomy-Based Frequency (ABF) Allocations on Early Performance Outcomes in MED-EL Cochlear Implant Recipients
Brief Title: Impact of Anatomy-Based Cochlear Implant Programming on Early Performance
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: US2401 MED-EL ABF
Record Dates: First submitted 2024-12-05; First posted 2024-12-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Unilateral; Cochlear Implants; Hearing Loss, Sensorineural; Single-Sided Deafness (SSD); Asymmetric Hearing Loss
Keywords: cochlear implant; Single-Sided Deafness
MeSH Terms: conditions — Hearing Loss, Unilateral; Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded to each of the frequency settings they are utilizing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Default Clinical Frequency Setting (Active Comparator): The audio processor frequency setting will be programmed based on current frequency defaults in the clinical programming software
  Interventions: Device: Programming of cochlear implant audio processor frequency settings
- Default Anatomy-Based Fitting (Active Comparator): The audio processor frequency setting will be programmed based on current anatomy-based fitting frequency defaults in the clinical programming software
  Interventions: Device: Programming of cochlear implant audio processor frequency settings
- Experimental Anatomy-Based Fitting 1 (Experimental): The audio processor frequency setting will be programmed using experimental settings for anatomy-based fitting using individual anatomical information obtained from analysis of post-operative imaging.
  Interventions: Device: Programming of cochlear implant audio processor frequency settings
- Experimental Anatomy-Based Fitting 2 (Experimental): The audio processor frequency setting will be programmed with experimental settings for anatomy-based fitting using individual anatomical information obtained from analysis of post-operative imaging.
  Interventions: Device: Programming of cochlear implant audio processor frequency settings

INTERVENTIONS:
Device: Programming of cochlear implant audio processor frequency settings — Cochlear implant audio processor frequency settings will be adjusted within the clinical programming software
  Other Names: anatomy-based fitting

SUMMARY:
The purpose of this study is to evaluate the impact of different audio processor frequency settings on performance outcomes in new cochlear implant users using electric-only stimulation in the implanted ear with normal hearing to moderately severe hearing loss in the opposite ear.

DETAILED DESCRIPTION:
Participants will be randomized into a starting frequency setting at device activation or shortly after device activation for the first three months of device use. After 3 months listening experience, participants will be randomized into different frequency settings and tested before and after a period of listening experience. Participant outcomes for each of the multiple frequency settings will be evaluated using standard clinical speech testing and through questionnaires designed to capture information about patient sound quality and quality of life.

ELIGIBILITY:
* At least 18 years of age
* Is a cochlear implant candidate as deemed by the participating center
* Implanted (or to be implanted) unilaterally with a MED-EL cochlear implant with moderately severe or better acoustic hearing in the contralateral ear.
* For patients who are already implanted, device activation must have occurred within 2 weeks of enrollment
* Patients with moderate contralateral hearing loss or greater must utilize a hearing aid in the contralateral ear.
* Programmed with electric-only stimulation in the implanted ear
* The ear to be implanted, acoustic hearing thresholds must be no better than 50 dBHL at 250 Hz and 65 dBHL at 500 Hz
* Post-operative CT scan allows for completion of OTOPLAN analysis
* ABF settings possible at defaults in clinical programming software
* Minimum of 10 active electrodes at activation
* Programmed using a Fine Structure coding strategy
* English is the primary language
* Willing and able to comply with all scheduled procedures as defined in the protocol

Exclusion Criteria:

* Subjects who do not meet one or more of the above-mentioned inclusion criteria are excluded from the study
* Subjects required to use a hearing aid per inclusion criteria who stop use of a hearing aid in the contralateral ear will be withdrawn at the time of discontinued hearing aid use
* Subjects who receive a cochlear implant in the contralateral ear prior to the 12-month interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Percent correct on AzBio Sentences in Noise | 3 to 7 months
  The AzBio sentence test, consisting of lists of 20 sentences spoken by male and female talkers, will be tested in noise in three spatial listening conditions with after listening experience with each frequency setting. Listening conditions include co-located presentation of the target and noise, target presented with noise to the implanted ear, and target presented with noise to the opposite acoustic hearing ear. Outcomes will be reported as percent correct (%).
Cochlear Implant Quality of Life - 35 Profile (CIQoL 35) | Enrollment to 7 months
  Subjects will complete a 35-item questionnaire with a total score ranging from 0-100% (higher score indicates a higher level of functional ability with a cochlear implant) regarding their subjective listening experience in 6 domains: communication, emotional, entertainment, environment, listening effort, social.

SECONDARY OUTCOMES:
Post-operative Audiogram | Enrollment and 12 months
  Unaided pure-tone audiometric thresholds will be tested for both ears. For patients with moderate to moderately severe hearing loss in the unimplanted ear, thresholds will also be tested in the best-aided condition.
Percent Correct on Az Bio Sentences in Noise | 12 months
  The AzBio sentence test, consisting of lists of 20 sentences spoken by male and female talkers, will be tested in noise in three spatial listening conditions with after listening experience with each frequency setting. Listening conditions include co-located presentation of the target and noise, target presented with noise to the implanted ear, and target presented with noise to the opposite acoustic hearing ear. Outcomes will be reported as percent correct (%).
Percent Correct on Consonant Nucleus Consonant (CNC) Words | 3 to 12 months
  The CNC test, consisting of 50 words scored as percent correct, will be tested in quiet after listening experience with each frequency setting for the implanted ear alone.
Subjective feedback questionnaire | Enrollment to 12 months
  Subjects will complete a non-validated subjective questionnaire assessing their perceptual sound quality prior to and after listening experience with different frequency settings. The questionnaire utilizes multiple choice questions, a 5-point Likert scale, and open-ended questions intended to collect subject feedback.
Psychoacoustic Testing of Sound Quality and Preference | 7 months
  Subjects will listen to speech and non-speech sounds will rate the quality of each sound on a 6-point Likert scale using different frequency settings. Subjects will then be asked to rank the different frequency settings relative to each other for quality and preference.
Cochlear Implant Quality of Life- 35 Profile (CIQoL35) | 12 months
  Subjects will complete a 35-item questionnaire with a total score ranging from 0-100% (higher score indicates a higher level of functional ability with a cochlear implant) regarding their subjective listening experience in 6 domains: communication, emotional, entertainment, environment, listening effort, social.
Decisional Regret Scale | 3 to 12 months
  A validated questionnaire using a 5-point Likert scale to assess decisional regret after cochlear implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Katelyn Glassman, AuD, Principal Investigator — Med-El Corporation
Locations (3):
- United States (3):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of North Carolina, Chapel Hill, North Carolina
  - MED-EL Corporation, Durham, North Carolina

REFERENCES:
- [Background] Shannon CM, Schvartz-Leyzac KC, Dubno JR, McRackan TR. Determinants of Cochlear Implant Satisfaction and Decisional Regret in Adult Cochlear Implant Users. Otol Neurotol. 2023 Dec 1;44(10):e722-e729. doi: 10.1097/MAO.0000000000004028. Epub 2023 Oct 19. PMID 37853774
- [Background] Sturm JJ, Ma C, McRackan TR, Schvartz-Leyzac KC. Frequency-to-Place Mismatch Impacts Cochlear Implant Quality of Life, But Not Speech Recognition. Laryngoscope. 2024 Jun;134(6):2898-2905. doi: 10.1002/lary.31264. Epub 2024 Jan 12. PMID 38214299
- [Background] Kurz A, Herrmann D, Muller-Graff FT, Voelker J, Hackenberg S, Rak K. Anatomy-based fitting improves speech perception in noise for cochlear implant recipients with single-sided deafness. Eur Arch Otorhinolaryngol. 2025 Jan;282(1):467-479. doi: 10.1007/s00405-024-08984-4. Epub 2024 Sep 19. PMID 39299967
- [Background] Fan X, Yang T, Fan Y, Song W, Gu W, Lu X, Chen Y, Chen X. Hearing outcomes following cochlear implantation with anatomic or default frequency mapping in postlingual deafness adults. Eur Arch Otorhinolaryngol. 2024 Feb;281(2):719-729. doi: 10.1007/s00405-023-08151-1. Epub 2023 Aug 7. PMID 37548704
- [Background] Kurz A, Herrmann D, Hagen R, Rak K. Using Anatomy-Based Fitting to Reduce Frequency-to-Place Mismatch in Experienced Bilateral Cochlear Implant Users: A Promising Concept. J Pers Med. 2023 Jul 8;13(7):1109. doi: 10.3390/jpm13071109. PMID 37511722
- [Background] Creff G, Lambert C, Coudert P, Pean V, Laurent S, Godey B. Comparison of Tonotopic and Default Frequency Fitting for Speech Understanding in Noise in New Cochlear Implantees: A Prospective, Randomized, Double-Blind, Cross-Over Study. Ear Hear. 2024 Jan-Feb 01;45(1):35-52. doi: 10.1097/AUD.0000000000001423. Epub 2023 Oct 12. PMID 37823850
- [Background] Dillon MT, Canfarotta MW, Buss E, Rooth MA, Richter ME, Overton AB, Roth NE, Dillon SM, Raymond JH, Young A, Pearson AC, Davis AG, Dedmon MM, Brown KD, O'Connell BP. Influence of Electric Frequency-to-Place Mismatches on the Early Speech Recognition Outcomes for Electric-Acoustic Stimulation Users. Am J Audiol. 2023 Mar;32(1):251-260. doi: 10.1044/2022_AJA-21-00254. Epub 2023 Feb 17. PMID 36800505
- [Background] Tan CT, Martin B, Svirsky MA. Pitch Matching between Electrical Stimulation of a Cochlear Implant and Acoustic Stimuli Presented to a Contralateral Ear with Residual Hearing. J Am Acad Audiol. 2017 Mar;28(3):187-199. doi: 10.3766/jaaa.15063. PMID 28277210
- [Background] Svirsky MA, Fitzgerald MB, Sagi E, Glassman EK. Bilateral cochlear implants with large asymmetries in electrode insertion depth: implications for the study of auditory plasticity. Acta Otolaryngol. 2015 Apr;135(4):354-63. doi: 10.3109/00016489.2014.1002052. Epub 2015 Feb 26. PMID 25719506
- [Background] Mertens G, Van de Heyning P, Vanderveken O, Topsakal V, Van Rompaey V. The smaller the frequency-to-place mismatch the better the hearing outcomes in cochlear implant recipients? Eur Arch Otorhinolaryngol. 2022 Apr;279(4):1875-1883. doi: 10.1007/s00405-021-06899-y. Epub 2021 Jun 15. PMID 34131770
- [Background] Canfarotta MW, Dillon MT, Buss E, Pillsbury HC, Brown KD, O'Connell BP. Frequency-to-Place Mismatch: Characterizing Variability and the Influence on Speech Perception Outcomes in Cochlear Implant Recipients. Ear Hear. 2020 Sep/Oct;41(5):1349-1361. doi: 10.1097/AUD.0000000000000864. PMID 32205726
- [Background] Goupell MJ, Noble JH, Phatak SA, Kolberg E, Cleary M, Stakhovskaya OA, Jensen KK, Hoa M, Kim HJ, Bernstein JGW. Computed-Tomography Estimates of Interaural Mismatch in Insertion Depth and Scalar Location in Bilateral Cochlear-Implant Users. Otol Neurotol. 2022 Jul 1;43(6):666-675. doi: 10.1097/MAO.0000000000003538. PMID 35761459
- [Background] Fitzgerald MB, Prosolovich K, Tan CT, Glassman EK, Svirsky MA. Self-Selection of Frequency Tables with Bilateral Mismatches in an Acoustic Simulation of a Cochlear Implant. J Am Acad Audiol. 2017 May;28(5):385-394. doi: 10.3766/jaaa.15077. PMID 28534729
- [Background] Fitzgerald MB, Sagi E, Jackson M, Shapiro WH, Roland JT Jr, Waltzman SB, Svirsky MA. Reimplantation of hybrid cochlear implant users with a full-length electrode after loss of residual hearing. Otol Neurotol. 2008 Feb;29(2):168-73. doi: 10.1097/mao.0b013e31815c4875. PMID 18165793
- [Background] Shannon RV. The relative importance of amplitude, temporal, and spectral cues for cochlear implant processor design. Am J Audiol. 2002 Dec;11(2):124-7. doi: 10.1044/1059-0889(2002/013). PMID 12691223
- [Background] Fu QJ, Shannon RV. Effects of electrode configuration and frequency allocation on vowel recognition with the Nucleus-22 cochlear implant. Ear Hear. 1999 Aug;20(4):332-44. doi: 10.1097/00003446-199908000-00006. PMID 10466569
- [Background] Dorman MF, Loizou PC, Rainey D. Simulating the effect of cochlear-implant electrode insertion depth on speech understanding. J Acoust Soc Am. 1997 Nov;102(5 Pt 1):2993-6. doi: 10.1121/1.420354. PMID 9373986